CLINICAL TRIAL: NCT03612869
Title: Open-label, Single-arm, Multi-center Study of Intracerebral Administration of Adeno-associated Viral (AAV) Serotype rh.10 Carrying Human N-sulfoglucosamine Sulfohydrolase (SGSH) cDNA for Treatment of Mucopolysaccharidosis Type IIIA
Brief Title: Study of AAVrh10-h.SGSH Gene Therapy in Patients With Mucopolysaccharidosis Type IIIA (MPS IIIA)
Acronym: AAVance
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LYSOGENE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P4-SAF-302
Record Dates: First submitted 2018-07-04; First posted 2018-08-02 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Mucopolysaccharidosis Type IIIA
Keywords: MPS IIIA; Sanfilippo syndrome Type A; Mucopolysaccharidosis Type IIIA; Lysosomal Storage Disease
MeSH Terms: conditions — Mucopolysaccharidosis III; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AAV SGSH gene therapy (LYS-SAF302) (Experimental): One-time intracerebral administration of adeno-associated viral vector serotype rh10 containing the human N-sulfoglucosamine sulfohydrolase (SGSH) cDNA.
  Interventions: Drug: LYS-SAF302

INTERVENTIONS:
Drug: LYS-SAF302 — Treatment will involve direct injections of the investigational product into both sides of the brain through image-guided tracks, in a single neurosurgical session.
  Other Names: AAVrh10-h.SGSH

SUMMARY:
MPS IIIA is predominantly a central nervous system disease causing cognitive disability, progressive loss of acquired skills, behavioral and sleep disturbance. LYS-SAF302 is a gene therapy which is intended to deliver a functional copy of the SGSH gene to the brain. This is a phase 2-3 study to assess the efficacy in improving or stabilizing the neurodevelopmental state of MPS IIIA patients.

DETAILED DESCRIPTION:
The study is interventional, single arm and multi-center. Evolution under treatment will be compared to expected natural evolution based on natural history studies.

ELIGIBILITY:
Inclusion Criteria:

* Documented MPS IIIA diagnosis based on genotyping confirming the SGSH gene mutations
* Cognitive DQ score on BSID-III: 50% and above

Exclusion Criteria:

* Homozygous for the S298P mutation or non-classical severe form of MPS IIIA, based on investigator's judgement.
* Participation in another gene or cell therapy clinical trial.
* Past use of SGSH enzyme replacement therapy for a period exceeding 3 months. A washout period of at least 2 months is required prior to screening.
* Current participation in a clinical trial of another investigational medicinal product.
* History of bleeding disorder or current use of medications that, in the opinion of the investigator, place them at risk of bleeding following surgery.
* Any condition that would contraindicate treatment with immunosuppressants such as tacrolimus, mycophenolate mofetil or steroids.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in development quotient (DQ), compared to regression reported in natural history studies | Month 6, 12, 18, 24
  Development Quotient will be measured for each patient using one of two standard instruments, the Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) or the Kaufman Assessment Battery for Children, Second Edition (KABC-II), based on age and ability range. The development quotient (DQ) is a means to express a neurodevelopmental/cognitive delay which is computed as a ratio and expressed as a percentage using the development age (DA) score divided by the age at testing ([development age score/chronological age] × 100; range: 0 - 100, where high values are desirable).

SECONDARY OUTCOMES:
Change from baseline in the total adaptive behavior composite standard score as measured by the expanded interview Vineland Adaptive Behavior Scales (VABS-II) | Month 6, 12, 18, 24
  The Vineland Adaptive Behavior Scales VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. The VABS-II is a norm-based instrument, where the child's adaptive functioning is compared to that of others his or her age. The total adaptive behavior composite score describe the child's functioning. The normative mean score is 100 (normative standard deviation is 15). Higher scores indicate better functioning.
Change in sleep pattern as measured by the Childrens Sleep Habits Questionnaire (CSHQ) | Month 6, 12, 18, 24
  The Children's Sleep habits Questionnaire (CSHQ) measures sleep habits and behavioral sleep disorders in preschool and school-aged children. The abbreviated CSHQ is a 23-item multiple-choice questionnaire that is summed into 8 subscales (bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night waking, parasomnias, sleep-disordered breathing, and daytime sleepiness) and a CSHQ total score, where higher scores reflect greater disturbance in sleep pattern. Scores will be compared to scores from the Natural History control group, using the same tool and same timepoints.
Change from baseline in patient quality of life using the Infant and Toddler Quality of Life (ITQOL) questionnaire | Month 12, 24
  The 47-item ITQOL questionnaire assesses physical, mental, and social well-being of the child and the quality of life of parent/caregiver. Scores range from 0 to 100, where higher scores reflect better quality of life. Change in score from baseline will be compared to scores from the Natural History control group, using the same tool and same timepoints.
Change from baseline in parent quality of life, using the Parenting Stress Index, 4th Edition (PSI-4) | Month 12, 24
  The 36-item questionnaire (PSI-4) is used to identify parent-child problem areas, measuring 3 main domains (parental distress, parent-child dysfunctional interaction, and difficult child), which all combined form a total stress score. Higher scores reflect a higher level of stress. Change in score from baseline will be compared to scores from the Natural History control group, using the same tool and same timepoints.
Change from baseline in total cortical grey matter volume and white matter volume on MRI | Month 12, 24
  The change from baseline in grey matter and white matter volume will be assessed by magnetic resonance imaging (MRI)
Incidence and severity of treatment-emergent adverse events and serious adverse events throughout the study | Month 24
  Descriptive summary tables for the surgical period, the evaluation period, and the follow-up period will be provided.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - CHOC Children's, Orange, California
  - University of Minnesota, Minneapolis, Minnesota
  - Weill Cornell Medical College, New York, New York
  - Baylor college of medicine / Texas children's hospital, Houston, Texas
- Armand Trousseau Public Hospital, Paris, France
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Amsterdam UMC, Amsterdam, Netherlands
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tardieu M, Zerah M, Husson B, de Bournonville S, Deiva K, Adamsbaum C, Vincent F, Hocquemiller M, Broissand C, Furlan V, Ballabio A, Fraldi A, Crystal RG, Baugnon T, Roujeau T, Heard JM, Danos O. Intracerebral administration of adeno-associated viral vector serotype rh.10 carrying human SGSH and SUMF1 cDNAs in children with mucopolysaccharidosis type IIIA disease: results of a phase I/II trial. Hum Gene Ther. 2014 Jun;25(6):506-16. doi: 10.1089/hum.2013.238. Epub 2014 May 5. PMID 24524415